CLINICAL TRIAL: NCT00794404
Title: Evaluation of Power Doppler US Technique for the Diagnosis of Spondylarthropathy in Patients With Uncertain Diagnosis Consulting for Clinical Symptoms Suggestive of Spondylarthropathy
Brief Title: Evaluation of Power Doppler US Technique for the Diagnosis of Spondylarthropathy
Acronym: EchoSpA
Status: Completed | Type: Observational
Sponsor: Dr Maria-Atonietta D'AGOSTINO (Other)
Collaborators: Groupe Français d'Etude Génétique des Spondylarthropathies (Other); French Society of Rheumatology (Other)
Responsible Party: Sponsor-Investigator, Dr Maria-Atonietta D'AGOSTINO, PU-PH, Groupe Français d'Etude Génétique des Spondylarthropathies
Organization: Groupe Français d'Etude Génétique des Spondylarthropathies (Other)
Other Study IDs: GESPA
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2008-11

CONDITIONS: Spondylarthropathy; Ankylosing Spondyloarthitis; Spondyloarthritis
MeSH Terms: conditions — Spondylarthropathies; Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the interest of enthesis sonography for the diagnosis of spondylarthritis, in patients with uncertain diagnosis consulting for clinical symptoms suggestive of spondylarthritis

DETAILED DESCRIPTION:
Spondylarthritis (SPA) are the second most frequent inflammatory rheumatic disorders and, because it starts early in life and has a chronic progressive course, the impact of this disease on health resources and patient's life quality can be important. Because the characteritic signs of SPA, like radiological evidence of sacro-iliitis, appear late in time, the lag time between the onset first signs of SPA for the patient and the confirmed diagnosis can be very long (up to 8 years). Previous studies proved that patients who are affected by SPA are showing abnormal vascularization of peripheral enthesis more frequently than patients affected by other rheumatic diseases. Ultrasonography in B mode combined with power Doppler (PDUS) is a non invasive and highly sensitive toll which can detect enthesitis and abnormal vsacularization even for the patients who are not showing yet the evidence of SPA's symptomatology. Using PDUS as a early diagnosis tool could lead to the improvement of diagnostic procedures and therapeutic management of SpA and reduce the cost of diagnosis for patient and health insurances.

ELIGIBILITY:
Inclusion Criteria:

* patients < 50 years old, consulting for spinal inflammatory symptoms > 3 months duration
* patients consulting for arthritis or tenderness joints > 3 months duration
* patients < 50 years old consulting for enthesitis or dactylitis > 3 months duration
* patients with uveitis and HLA-B27 positivity
* relatives of SpA patients consulting for symptoms suggestive of SpA

Exclusion Criteria:

* patient with confirmed diagnosis of rheumatic disease (included SpA)
* patient protected by law (patient <18 years old, pregnant woman)
* patient who can't atempt the RMI
* patient who will have difficulties to complete the two years of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a symptomatology which can lead to a SPA diagnosis but with no confirmed diagnosis yet for any rheumatic didease.
Sampling Method: Non-Probability Sample
Enrollment: 489 (Actual)
Dates: Start 2004-12; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D'AGOSTINO Maria-Antonietta, MCUPH, Principal Investigator — Ambroise Paré Hospital
Locations (6):
- France (6):
  - Ambroise Paré Hospital, Boulogne-Billancourt
  - Cavale Blanche Hospital, Brest
  - Cote de Nacre Hospital, Caen
  - South Hospital of Grenoble, Échirolles
  - Conception Hospital, Marseille
  - Nancy Brabois Hospital, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Devauchelle-Pensec V, D'Agostino MA, Marion J, Lapierre M, Jousse-Joulin S, Colin D, Chary-Valckenaere I, Marcelli C, Loeuille D, Aegerter P, Guis S, Gaudin P, Breban M, Saraux A; Study Group of Spondylarthritis. Computed tomography scanning facilitates the diagnosis of sacroiliitis in patients with suspected spondylarthritis: results of a prospective multicenter French cohort study. Arthritis Rheum. 2012 May;64(5):1412-9. doi: 10.1002/art.33466. PMID 22081446